CLINICAL TRIAL: NCT03646253
Title: Analysis of Four-fragment Fractures of the Proximal Humerus: the Interest of 2D and 3D Imagery and Inter- and Intra-observer Reproducibility
Acronym: REPROD-HUMERUS
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao005
Record Dates: First submitted 2018-08-07; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Reproducibility; Four Part Fracture; Proximal Humerus Fracture; Hertel's Criteria
Keywords: Proximal humerus fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with proximal humerus fracture
  Interventions: Other: Analysis of radiology (standard radiographies, 2D scan sections and 3D reconstructions)

INTERVENTIONS:
Other: Analysis of radiology (standard radiographies, 2D scan sections and 3D reconstructions)

SUMMARY:
Fractures of the proximal humerus are increasingly frequent, with numbers tripling between the 1970s and the 2000s. Among these fractures, those involving the tuberosities and also the anatomic neck are a therapeutic challenge. For this type of fracture (Neer's four-part fracture) the degree of displacement of the fracture needs to be understood in order to provide suitable treatment and apprehend the risks in its evolution. There is indeed, in this type of fracture, a risk of humeral head ischaemia, which will carry considerable weight in the therapy adopted.

The usual classifications, such as the AO or the Neer classification, have shown their limitations in terms of reproducibility and are not suitable for the prognostic assessment of these four-fragment fractures of the proximal humerus. The radiographic parameters described by Hertel in 2004, on the other hand, seem to be far more relevant to routine clinical practice.

The use of the scanner to improve reproducibility of the classification of these proximal humerus fractures is still controversial. The scanner is the rule to guide therapeutic strategy for complex fractures, although the reproducibility of the different assessment criteria has never been studied.

DETAILED DESCRIPTION:
The aims of the present study were firstly to analyse inter-observer and intra-observer reproducibility for the different criteria proposed by Hertel, using three types of imagery (standard radiographies, 2D and 3D scans) and secondly to assess the relevance of the use of the scanner to improve reproducibility

ELIGIBILITY:
Inclusion Criteria:

* Proximal humerus fracture
* standard radiographs, a 2D scan with axial, sagittal and coronal sections, and high-resolution 3D reconstructions performed in emergency settings when the patient arrived in the care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Inter-rater reproducibility concerning displacement of the humeral head on the frontal plane for 3D reconstructions | Day 0
  Displacement of the humeral head on the frontal plane evaluated in "not displaced", "varus" or "valgus".
  Assessment of inter-rater reproductibility for displacement of the humeral head on the frontal plane using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning displacement of the humeral head on the sagittal plane for 3D reconstructions | Day 0
  Displacement of the humeral head on the sagittal plane evaluated in "not displaced", "angle more than 20 degrees" or "angle less than 20 degrees".
  Assessment of inter-rater reproductibility for displacement of the humeral head on the sagittal plane using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning humeral head split for 3D reconstructions | Day 0
  Humeral head split evaluated in "presence" or "absence". Assessment of inter-rater reproductibility for humeral head split using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning calcar comminution for 3D reconstructions | Day 0
  Calcar comminution evaluated in "presence" or "absence". Assessment of inter-rater reproductibility for calcar comminution using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning medial hinge for 3D reconstructions | Day 0
  Medial hinge evaluated in "presence" or "absence". Assessment of inter-rater reproductibility for medial hinge using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning length of metaphyseal extension for 3D reconstructions | Day 0
  Length of metaphyseal extension evaluated in "less than 8 mm" or "more than 8 mm".
  Assessment of inter-rater reproductibility for length of metaphyseal extension using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning displacement of the greater tuberosity for 3D reconstructions | Day 0
  Displacement of the greater tuberosity evaluated in "not displaced", "more than 5 mm" or "less than 5 mm".
  Assessment of inter-rater reproductibility for displacement of the greater tuberosity using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.
Inter-rater reproducibility concerning displacement of the lesser tuberosity for 3D reconstructions | Day 0
  Displacement of the lesser tuberosity evaluated in "not displaced", "more than 5 mm" or "less than 5 mm".
  Assessment of inter-rater reproductibility for displacement of the lesser tuberosity using Cohen's Kappa coefficient. A Kappa coefficient comprised between 0.00 and 0.20 significate a very poor agreement, between 0.21 and 0.40 significate a poor agreement, between 0.41 and 0.60 significate a moderate agreement, between 0.61 and 0.80 significate a satisfactory agreement and between 0.81 and 1.00 significate an excellent agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Ohl X, Mangin P, Barbe C, Brun V, Nerot C, Sirveaux F. Analysis of four-fragment fractures of the proximal humerus: the interest of 2D and 3D imagery and inter- and intra-observer reproducibility. Eur J Orthop Surg Traumatol. 2017 Apr;27(3):295-299. doi: 10.1007/s00590-017-1911-2. Epub 2017 Jan 24. PMID 28120098